CLINICAL TRIAL: NCT05714969
Title: A Phase 2b, Multicenter, Randomized, Double-blind Study of Safety and Efficacy of TAK-755 (rADAMTS13) With Minimal to No Plasma Exchange (PEX) in the Treatment of Immune-mediated Thrombotic Thrombocytopenic Purpura (iTTP)
Brief Title: A Study of TAK-755 (rADAMTS13) With Little to No Plasma Exchange (PEX) Treatment in Adults With Immune-mediated Thrombotic Thrombocytopenic Purpura (iTTP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-755-2001; 2023-507787-39-00 (EU CTIS Number)
Record Dates: First submitted 2023-01-24; First posted 2023-02-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
Keywords: Drug Therapy; Immune-mediated Thrombotic Thrombocytopenic Purpura (iTTP)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — ADAMTS13 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is double-blind, randomization and Part 2 is open-label, single-arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: TAK-755 Dose 1 in Acute Phase and Dose 2 in Post-acute Phase (Experimental): TAK-755 Dose 1, IV infusion, in the acute phase until clinical response is achieved. All participants achieving clinical response will receive TAK-755 at Dose 2, for up to 6 weeks during the post-acute phase.
  Interventions: Biological: TAK-755
- Part 1: TAK-755 Dose 2 in Both Acute and Post-Acute Phase (Experimental): TAK-755 Dose 2, IV infusion, in the acute phase until clinical response is achieved. All participants achieving clinical response will receive TAK-755 at Dose 2, for up to 6 weeks during the post-acute phase.
  Interventions: Biological: TAK-755
- Part 2: TAK-755 Dose 3 in Acute Phase and Dose 2 in Post-acute Phase (Experimental): TAK-755 Dose 3, IV infusion, in the acute phase until 48-hour platelet response is achieved. All participants achieving platelet response will receive TAK-755 at Dose 2, 4 times per week for Week 1 and 3 times per week for Week 2 and 3 during the post-acute phase based on investigator judgement as high-risk for developing iTTP recurrence.
  Interventions: Biological: TAK-755

INTERVENTIONS:
Biological: TAK-755 — TAK-755 IV infusion
  Other Names: rADAMTS13; recombinant ADAMTS13; SHP-655; BAX 930

SUMMARY:
This is a study of TAK-755 in adults with immune-mediated thrombotic thrombocytopenic purpura (iTTP). The main aim of this study is to determine the percentage of participants with a clinical (Part 1) or platelet (Part 2) response without plasma exchange during the study. Participants who have an acute attack of iTTP will receive TAK-755 and immunosuppressive therapy during their stay at the hospital until they achieve a clinical response in Part 1 or platelet response in Part 2. Participants will also be treated with TAK-755 for an additional time of up to 6 weeks after the acute phase. In total, participants will stay in the study for approximately 3 months.

DETAILED DESCRIPTION:
This study consists of 2-parts. Part 1 is a double-blind, randomized study in which participants were randomized 1:1, in a blinded fashion, into 2 TAK-755 dose groups. Part 1, randomization was stratified based on whether the participant had received pre-study PEX and on the participant's Glasgow Coma Scale. Part 2 is an open-label study in which participants with iTTP experiencing an acute iTTP episode will be enrolled and assigned to a single-arm treatment.

ELIGIBILITY:
Key Inclusion Criteria (Part 1 and Part 2)

1. Participant must provide a signed informed consent form. A fully recognized proxy may be used per local laws for participants unable to provide consent.
2. Participant is 18 years or older at time of screening.
3. Participant has been diagnosed with de novo or relapsed iTTP.
4. Participant must be willing to fully comply with study procedures and requirements.
5. Female participants of childbearing potential must present with a negative pregnancy test and agree to employ highly effective birth control measures for duration of study. Sexually active male participants must agree to use an effective method of contraception for the duration of the study.

Key Exclusion Criteria (Part 1 and Part 2)

1. Participant has received more than 2 pre-study PEX prior to randomization in Part 1 or first dose of investigational product in Part 2.
2. Participant has been diagnosed with cTTP or another cause of thrombotic microangiopathy (TMA).
3. Participant has been exposed to another investigational product within 30 days prior to enrollment or is scheduled to participate in another clinical study involving investigational product or investigational device during the course of the study.
4. Participant has received caplacizumab within 30 days prior to study enrollment.
5. Participant has had a previous iTTP event within the past 30 days.
6. Participant is positive for human immunodeficiency virus (HIV) with unstable disease or cluster of differentiation (CD)4+ count ≤200 cells/mm^3 within 3 months of screening.
7. Participant has condition of severe immunodeficiency.
8. Participant has a severe systemic acute infection.
9. Participant has another underlying progressive fatal disease and/or life expectancy <3 months.
10. Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures.
11. Participant is pregnant or lactating.
12. Participant has any condition in which methylprednisolone or other steroid equivalent is contraindicated as per prescribing information.
13. Participant has known life-threatening hypersensitivity reaction, including anaphylaxis, to the parent molecule ADAMTS13, Chinese hamster ovary (CHO) cell proteins, or other constituents of TAK-755.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-06-11 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Event of Special Interest (AESIs) After Receiving any Dose of Investigational Product (IP) | Through study completion, approximately 12 weeks
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. SAE: Signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event. Adverse events of special interest include major thrombotic events and treatment-related bleeding events.

SECONDARY OUTCOMES:
Part 1: Achievement of Clinical Response Without On-Study Plasma Exchange (PEX) | Through study completion, approximately 12 weeks
  Clinical response is defined as normalization of platelets and no clinical evidence of new or progressive ischemic organ injury. Normalization of platelets: First occurrence of normal platelet count (greater than or equal to [>=]150,000/microliter [mcL]) that is followed by a confirmatory platelet count of >=150,000/mcL and a lactate dehydrogenase (LDH) <1.5×upper limit of normal (ULN) at 48±12 hours after the first occurrence.
Part 2: Achievement of Platelet Response Without On-Study Plasma Exchange (PEX) | Through study completion, approximately 12 weeks
  Platelet response is defined as first occurrence of normal platelet count (>=150,000/mcL) that is followed by a confirmatory platelet count of >=150,000/mcL at 48±12 hours after the first occurrence.
Part 1: Achievement of Clinical Response With Zero or Minimal on-Study PEX | Through study completion, approximately 12 weeks
  The number of PEX administered considered Zero when no PEX is administered and considered Minimal when 1 to 3 PEX are administered.
Part 2: Achievement of Platelet Response With Zero or Minimal on-Study PEX | Through study completion, approximately 12 weeks
  The number of PEX administered considered Zero when no PEX is administered and considered Minimal when 1 to 3 PEX are administered.
Part 1: Achievement of Clinical Response Overall | Through study completion, approximately 12 weeks
  Overall indicates clinical response regardless of whether on-study PEX is administered, or the number of PEX administered.
Part 2: Achievement of Platelet Response Overall | Through study completion, approximately 12 weeks
  Overall indicates platelet response regardless of whether on-study PEX is administered, or the number of PEX administered.
Part 1: Time to Clinical Response (Acute Phase) | Through study completion, approximately 12 weeks
Part 2: Time to Platelet Response (Acute Phase) | Through study completion, approximately 12 weeks
Part 1: Occurrence of Refractoriness (Acute Phase) | Through study completion, approximately 12 weeks
Part 1: Time to First On-Study PEX in Participants who Achieved Clinical Response | Through study completion, approximately 12 weeks
Part 2: Time to First On-Study PEX in Participants who Achieved Platelet Response | Through study completion, approximately 12 weeks
Part 1: Number of Days of On-study PEX in Participants to Achieve Clinical Response (Acute Phase) | Through study completion, approximately 12 weeks
Part 2: Number of Days of On-study PEX in Participants to Achieve Platelet Response (Acute Phase) | Through study completion, approximately 12 weeks
Part 1: Total Volume of Plasma Administered (Acute Phase) to Achieve Clinical Response | Through study completion, approximately 12 weeks
Part 2: Total Volume of Plasma Administered (Acute Phase) to Achieve Platelet Response | Through study completion, approximately 12 weeks
Part 1: Occurrence of Treatment Failure | Through study completion, approximately 12 weeks
  Treatment failure is defined as failure to achieve clinical response, or experience iTTP recurrence.
Part 2: Occurrence of Treatment Failure | Through study completion, approximately 12 weeks
  Treatment failure is defined as failure to achieve platelet response, or experience iTTP recurrence.
Part 1: Occurrence of Immune-Mediated Thrombotic Thrombocytopenic Purpura (iTTP) Recurrence (Following Clinical Response), Exacerbation, or Relapse (Post-acute Phase) | Through study completion, approximately 12 weeks
  iTTP recurrence comprised of exacerbation or relapse. Clinical exacerbation: Occurs <30 days after achieving initial clinical response (i.e., before clinical remission) and recurrent thrombocytopenia (platelet levels <150,000/μL), with or without clinical evidence of new or progressive ischemic organ damage, requiring daily PEX or rescue therapy. Clinical relapses: Occurs >=30 days after achieving initial clinical response (i.e., after clinical remission) and recurrent thrombocytopenia (platelet levels <150,000/μL), with or without clinical evidence of new or progressive ischemic organ damage, requiring daily PEX or rescue therapy.
Part 2: Occurrence of iTTP Recurrence (Following Platelet Response), Exacerbation, or Relapse (Post-acute Phase) | Through study completion, approximately 12 weeks
  iTTP recurrence comprised of exacerbation or relapse. Clinical exacerbation: Occurs <30 days after achieving initial platelet response (i.e., before clinical remission) and recurrent thrombocytopenia (platelet levels <150,000/μL), with or without clinical evidence of new or progressive ischemic organ damage, requiring daily PEX or rescue therapy. Clinical relapses: Occurs >=30 days after achieving initial platelet response (i.e., after clinical remission) and recurrent thrombocytopenia (platelet levels <150,000/μL), with or without clinical evidence of new or progressive ischemic organ damage, requiring daily PEX or rescue therapy.
Part 1: Time to iTTP Recurrence (Following Clinical Response), Exacerbation, or Relapse | Through study completion, approximately 12 weeks
Part 2: Time to iTTP Recurrence (Following Platelet Response), Exacerbation, or Relapse | Through study completion, approximately 12 weeks
Part 1: Occurrence of Any One of the Following Events: Clinical Recurrence (Following Clinical Response), iTTP-Related Death, or Major Thrombotic Event From Time of First IP Administration Through Study Completion | Through study completion, approximately 12 weeks
Part 2: Occurrence of Any One of the Following Events: Clinical Recurrence (Following Platelet Response), iTTP-Related Death, or Major Thrombotic Event From Time of First IP Administration Through Study Completion | Through study completion, approximately 12 weeks
Part 1: Time to Occurrence of Any One of the Following Events: Clinical Recurrence (Following Clinical Response), iTTP-Related Death, or Major Thrombotic Event From Time of First IP Administration Through Study Completion | Through study completion, approximately 12 weeks
Part 2: Time to Occurrence of Any One of the Following Events: Clinical Recurrence (Following Platelet Response), iTTP-Related Death, or Major Thrombotic Event From Time of First IP Administration Through Study Completion | Through study completion, approximately 12 weeks
Part 1: Change From Baseline in Lactate Dehydrogenase [LDH] Levels at Clinical Response and Study Completion | Through study completion, approximately 12 weeks
Part 2: Change From Baseline in LDH Levels at Platelet Response and Study Completion | Through study completion, approximately 12 weeks
Part 1: Change From Baseline in Troponin Levels at Clinical Response and Study Completion | Through study completion, approximately 12 weeks
Part 2: Change From Baseline in Troponin Levels at Platelet Response and Study Completion | Through study completion, approximately 12 weeks
Part 1: Achievement of Clinical Remission | Through study completion, approximately 12 weeks
  Clinical remission is defined as achieving clinical response and no recurrence for >=30 days.
Part 2: Achievement of Clinical Remission | Through study completion, approximately 12 weeks
  Clinical remission is defined as achieving platelet response and no recurrence for >=30 days.
Part 1 and 2: A Disintegrin and Metalloproteinase With Thrombospondin Motifs 13 (ADAMTS13) Antigen Level Resulting From TAK-755 Administration in Acute and Post-Acute Phases | Through study completion, approximately 12 weeks
Part 1 and 2: ADAMTS13 Activity Level Resulting From TAK-755 Administration in Acute and Post-Acute Phases | Through study completion, approximately 12 weeks
Part 1: Von Willebrand Factor (VWF) Antigen Level Resulting From TAK-755 Administration in Acute and Post-Acute Phases | Through study completion, approximately 12 weeks
Part 1: VWF Activity Level Resulting From TAK-755 Administration in Acute and Post-Acute Phases | Through study completion, approximately 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- United States (12):
  - University of Florida - Shands, Gainesville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Clinical Research Unit, Minneapolis, Minnesota
  - Rutgers University, New Brunswick, New Jersey
  - Weill Cornell, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Leo Jenkins Cancer Center/ECU School of Medicine, Greenville, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Versiti Wisconsin, Inc., Milwaukee, Wisconsin
- AKH - Medizinische Universitat Wien, Vienna, Austria
- General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki, Greece
- Italy (2):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino
- Spain (4):
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - University College London Hospital, London, Greater London
  - Royal Liverpool University Hospital, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: NOTE: IPD Sharing Time Frame has not been entered.
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/f5b44c8ac8e8425f?idFilter=%5B%22TAK-755-2001%22%5D